CLINICAL TRIAL: NCT03430960
Title: Defense and Veterans Pain Rating Scale (DVPRS)and Post Operative Survey Through a Bi-Directional Secure Mobile Messaging System - A Randomized Feasibility Study (mCare)
Brief Title: Post Operative Survey Through a Bi-Directional Secure Mobile Messaging System
Acronym: mCare
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Defense and Veterans Center for Integrative Pain Management (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 500249
Record Dates: First submitted 2017-11-28; First posted 2018-02-13 (Actual); Last update posted 2018-09-19 (Actual); Status verified 2018-09

CONDITIONS: Pain
Keywords: mCare; post surgery; mobile; healthcare; application
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A - Standard of Care (Other)
  Interventions: Other: Phone Call
- Group B - mCare group (Experimental)
  Interventions: Other: Mobile App Survey

INTERVENTIONS:
Other: Phone Call — Participants will be followed-up via phone call by Acute Pain Research Nurse
  Arms: Group A - Standard of Care
Other: Mobile App Survey — Participants will be followed-up via mCare mobile app
  Arms: Group B - mCare group

SUMMARY:
* Purpose The general purpose of this project is to assess the utility of the mCare application and MHCE (Mobile Healthcare Environment) system - a secure, mobile, smartphone app based platform - for same day surgery postoperative follow up of patients receiving peripheral nerve blocks.
* Research Design Randomized open-label study, comparing the satisfaction of the two groups with the method of follow up, which is either over the phone or via a mCare application. A separate group made up of nurses and physicians will have the opportunity to take a short anonymous survey to rank their opinion on the use of the smartphone application for patient feedback.

DETAILED DESCRIPTION:
The primary objective of the study is to evaluate the feasibility of the implementation of the mCare system for postoperative follow-up and querying of patients receiving peripheral nerve blocks during their perioperative care. The investigators intend to perform a randomized pilot study comparing mCare with the current standard of care. Participants will be randomized into 2 groups: a) standard of care groups and b) mCare group. In the standard of care group, the participants will be followed-up via a phone call by an Acute Pain Service (APS) nurse, according to current standards. During the past year there have been 375 calls made, 64 of which have not been answered (17%). In the mCare group participants will be followed-up via mCare application. 48 hours after discharge an APS nurse is going to call the participants in group a) and the mCare system will notify participants in group b) to answer follow-up questions about their pain and peripheral nerve block. If necessary (based on the follow-up algorithm), participants in either group will be contacted (via phone call or the app, depending on group assignment) 7 days after their surgery to assess resolution of the peripheral nerve block. At the end of follow-up, on postoperative day 8, each patient will be asked to complete the satisfaction and convenience surveys. 10 days after their surgery participants in the mCare group will complete the System Usability Survey (SUS).At the end of the study, APS nurses and medical providers will be asked to complete the satisfaction and convenience surveys, and follow-up response data will be summarized and analyzed. Our research question is whether the use of the mCare system would result in improved patient compliance, satisfaction, and convenience on both the patient and the provider side, while being at least as safe as the standard of care.

Research question 1: Does the use of mCare app improve postoperative follow-up response rate of patients receiving perioperative peripheral nerve blocks who are discharged the same day?

Research question 2: Does satisfaction, convenience and ease of use differ between the mCare system and current standards a) in the patient population and b) among health care providers?

The pain assessment tool adapted for the mCare app will be the Defense and Veterans Pain Rating Scale(DVPRS),which is a 6 item questionnaire for assessing current pain, average and worst pain over the last 24 hours, and physical and emotional function. The DVPRS has been validated at Walter Reed National Military Medical Center (WRNMMC), but the administration has been paper based during rounds by the Acute Pain Service.

The current standard for follow up with patients who receive regional anesthesia for same day surgery is that the APS nurse contacts them 48 hours after the procedure and asks about their pain, qualities and duration of the nerve block, and their satisfaction with the service. If the patient's answers make it necessary (e.g. the block doesn't wear off, the numbness still persists) then the APS nurse calls them again one week after the surgery. If the numbness still persists at that point, then the APS nurse escalates their case by informing the regional anesthesia provider who decides further steps.

In this study, the investigators intend to substitute the phone call by the APS nurse with the use of the mCare app. Our research question is whether the app is at least as safe as the standard of care, and at least as easy to use and convenient as the phone call.

ELIGIBILITY:
Inclusion Criteria:

* Male and female military health care beneficiaries age 18 and 89 years old
* Receive peripheral nerve block affecting their limb(s)
* Same day surgery
* Owns a personal cell phone with the following features:
* A 320 x 240 screen display resolution or greater
* ii. Text messaging capabilities
* iii. Data service capabilities
* iv. Service provided by either: AT&T, AllTel, Sprint, T-Mobile, or Verizon
* Ability to use their personal cell phone
* Ability to read and respond to a message in English as the app is only in English.
* Receives reliable cell phone service in their home.
* DEERS eligibility

Exclusion Criteria:

* Under age 18 and over 89 years old
* Non-English speaking-App will only be in English as this is an app developed just for this study.
* Active participation in other research studies involving mobile devices
* Inability to interact with a touch screen mobile device
* Receive Exparel(which is a pain medication drug they can receive during surgery since these patients will be called 48 hour post discharge)

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-06-16 (Actual); Primary Completion 2018-06-15 (Actual); Study Completion 2018-08-30 (Actual)

PRIMARY OUTCOMES:
Clinical Burden of Contact Method | 10 days
  This will be measured by comparing the proportion of patients who completed clinical measures at initial contact attempt and any contact attempt. The initial contact method is a phone call for the SOC group, and an initial text reminder for mCare group. Patients who do not respond to the initial contact attempt are subsequently re-contacted, which is a clinical burden.

SECONDARY OUTCOMES:
Participant-Reported Contact-Method Evaluations | 10 days
  A contact-method satisfaction survey asked participants the degree to which they were satisfied with their contact method (phone or mCare app) (1=not satisfied at all, 5=completely satisfied), whether they would like to use their respective contact method for follow-up after a future surgery (yes/no), and the degree to which the contact method was convenient (1=not convenient at all, 5=very convenient). An 8-item system usability survey was completed by mCare participants. Participants rated the degree to which they agreed with statements of app usability on a 5-point scale (1=strongly disagree, 5=strongly agree).
Nurse Satisfaction and Preferences | 10 days
  A 5-item nurse satisfaction survey assessed nurse satisfaction and preferences for each contact method. This included which method they gave more accurate information, was easier to understand and use, was more convenient, was safer, and preferred for post-surgical follow-up for regional anesthesia. Response options included: phone call, mCare, and both methods equally.

CONTACTS AND LOCATIONS:
Overall Officials: COL (ret) Chester C Buckenmaier, MD, Principal Investigator — Defense and Veterans Center for Integrative Pain Management
Locations (1):
- Walter Reed National Military Medical Center, Bethesda, Maryland, United States